CLINICAL TRIAL: NCT01685424
Title: Etoricoxib Prescribing Patterns and Adverse Events of Interest During Etoricoxib Treatment in UK Primary Care; an Updated Analysis
Brief Title: Etoricoxib Prescribing Patterns and Adverse Events of Interest in Primary Care in the United Kingdom (MK-0663-162 AM1)
Status: Completed | Type: Observational
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Other Study IDs: 0663-162; 7013.021 (Other: Study Identification Number); EMEA/H/A - 31/632 (Other: Regulatory identifier)
Record Dates: First submitted 2012-08-23; First posted 2012-09-14 (Estimated); Last update posted 2022-02-18 (Actual); Status verified 2022-02

CONDITIONS: Osteoarthritis; Rheumatoid Arthritis; Ankylosing Spondylitis; Gout; Arthritis
Keywords: Etoricoxib; ARCOXIA; Osteoarthritis; Rheumatoid Arthritis; Ankylosing Spondylitis; Gout; Arthritis
MeSH Terms: conditions — Osteoarthritis; Arthritis, Rheumatoid; Spondylitis, Ankylosing; Gout; Arthritis | interventions — Etoricoxib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Etoricoxib Prescription (Period 1): First Etoricoxib Prescription, Apr. 1, 2002 to Feb. 17, 2005
  Interventions: Drug: Etoricoxib
- Etoricoxib Prescription (Period 2): First Etoricoxib Prescription, Feb. 18, 2005 to Dec. 31, 2015
  Interventions: Drug: Etoricoxib
- Repeat Etoricoxib Prescription: One prescription during the Period 1 and, at least, one etoricoxib prescription during Period 2.
  Interventions: Drug: Etoricoxib

INTERVENTIONS:
Drug: Etoricoxib — As per routine clinical practice in the United Kingdom
  Other Names: ARCOXIA®)

SUMMARY:
This postmarketing study was conducted to describe prescribing patterns for etoricoxib (ARCOXIA®) in General Practice and describe the incidence of selected adverse events recorded in the United Kingdom (UK) Medicines and Health Care Products Regulatory Agency (MHRA) General Practice Research Database (GPRD).

ELIGIBILITY:
Inclusion Criteria:

* All patients in the MHRA's Full Feature GPRD (FF-GPRD) who have at least one electronic outpatient prescription record for etoricoxib issued by a General Practitioner during the period (April 1, 2002 to December 31, 2015) at the date of query execution against the FF-GPRD data warehouse.

Exclusion Criteria:

* Not registered in a GPRD-contributing practice that had continuously

collected data deemed to be 'up-to-standard' for research purposes from 1 April 2002 through to 31 December 2015.

* Never registered as a permanent patient of a General Practitioner in the practice
* Registration details were not acceptable (i.e. incomplete data or logically implausible dates)
* Not registered with a General Practitioner for at least 365 days before the date that the patient's first etoricoxib prescription was recorded in the GPRD

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All participants in the MHRA's Full Feature GPRD (FF-GPRD) who have at least one electronic outpatient prescription record for etoricoxib issued by a General Practitioner during the period (April 1, 2002 to December 31, 2015) at the date of query execution against the FF-GPRD data warehouse.
Sampling Method: Probability Sample
Enrollment: 79189 (Actual)
Dates: Start 2006-06-30 (Actual); Primary Completion 2015-03-01 (Actual); Study Completion 2015-03-01 (Actual)

PRIMARY OUTCOMES:
Dose of Initial Etoricoxib Prescription | At first prescription (during a time period up to 13.75 years)
Duration of Initial Etoricoxib Prescription | At first prescription (during a time period up to 13.75 years)
Participant's Baseline Characteristics (Demographics and Medical) | At first prescription (during a time period up to 13.75 years)
Incidence of Adverse Events of Special Interest Among Etoricoxib Users | During a time period up to 13.75 years

SECONDARY OUTCOMES:
"Off-label" use of Etoricoxib | At first prescription (during a time period up to 13.75 years)

REFERENCES:
- See also: EU PAS Register (EUPAS17526) — http://www.encepp.eu/encepp/viewResource.htm?id=19307